CLINICAL TRIAL: NCT07343934
Title: Phase 1 Study of huCART19-IL18-eDHFR Cells in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: huCART19-IL18-eDHFR Cells in Relapsed/Refractory Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Follicular Lymphoma Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 859859 (30425)
Record Dates: First submitted 2025-12-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Follicular Lymphoma
Keywords: Follicular Lymphoma; CAR T cells
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Dose Level -1 (DL-1) will only be explored if ≥ 2 Treatment Limited Toxicities occur at any time in DL1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - DL1 (Experimental): IV administration of a single flat dose of 7x10[6] huCART19-IL18-eDHFR cells. [18F]FP-TMP PET/CT scan.
  Interventions: Biological: huCART19-IL18-eDHFR cells; Drug: [18F]Fluoropropyl-Trimethoprim
- Arm A - DL-1 (Experimental): IV administration of a single flat dose of 3x10[6] huCART19-IL18-eDHFR cells. [18F]FP-TMP PET/CT scan.
  Interventions: Biological: huCART19-IL18-eDHFR cells; Drug: [18F]Fluoropropyl-Trimethoprim

INTERVENTIONS:
Biological: huCART19-IL18-eDHFR cells — Genetically modified autologous T cells engineered by co-transduction with two lentiviral vectors; one vector expressing a chimeric antigen receptor (CAR) targeting the CD19 antigen and human Interleukin 18 (IL-18), and a second vector expressing E.coli dihydrofolate reductase (eDHFR)
Drug: [18F]Fluoropropyl-Trimethoprim — Co-expression of eDHFR within huCART19-IL18 cells will allow the trafficking of the transduced CAR T cells to be visualized by PET/CT imaging using an investigational radiolabeled imaging agent [18F]Fluoropropyl-Trimethoprim (also known as [18F]FP-TMP).
  Other Names: [18F]FP-TMP

SUMMARY:
This is a phase 1, open-label study to evaluate the feasibility, safety and preliminary efficacy of huCART19-IL18-eDHFR cells administered in patients with relapsed or refractory follicular lymphoma. This study will be initiated as a single arm study (Treatment Arm A), which will evaluate the use of huCART19-IL18-eDHFR cells without prior lymphodepletion. In this Treatment Arm A, all subjects will receive a single flat dose of 7x10[6] huCART19-IL18-eDHFR cells (Dose Level 1; DL1). Additional treatment arms may also be introduced in the future, via subsequent amendment(s).

Co-expression of eDHFR within huCART19-IL18 cells will allow the trafficking of the transduced CAR T cells to be visualized by PET/CT imaging using an investigational radiolabeled imaging agent [18F]Fluoropropyl-Trimethoprim (also known as [18F]FP-TMP). The feasibility of using [18F]FP-TMP PET/CT imaging to detect and measure the eDHFR-expressing CAR T cells will be investigated, as well as its ability to provide insight into CAR T cell pharmacokinetics, biodistribution, and persistence.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Male or females age ≥ 18 years
3. Diagnosis of follicular lymphoma, grades 1-3A
4. Relapsed or refractory disease after at least 2 prior lines of systemic therapy as follows:

   1. Prior therapy must include an anti-CD20 monoclonal or bispecific antibody and an alkylating agent.
   2. Must have progressed within 2 years after second or higher line of therapy.
5. Documentation of CD19 expression on malignant cells by flow cytometry/IHC from a CLIA certified laboratory. Results must be within 6 months of physician-investigator confirmation of eligibility and after any intervening CD19 directed therapy since expression confirmed.
6. Patients with relapsed disease after prior allogeneic SCT must meet the following criteria:

   1. Have no active GVHD and require no immunosuppression
   2. Are more than 6 months from transplant at the time of physician-investigator confirmation of eligibility
7. Evidence of progressive disease within 12 weeks of physician-investigator confirmation of eligibility.
8. ECOG Performance Status that is either 0 or 1.
9. Adequate organ function defined as:

   1. Serum creatinine ≤ 1.5x ULN or estimated creatinine clearance ≥ 35 mL/min and not on dialysis
   2. ALT/AST ≤ 3 x ULN
   3. Direct bilirubin ≤ 2.0 mg/dl; for patients with Gilbert's syndrome direct bilirubin must be ≤ 3.0 mg/dl
   4. Left Ventricular Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
   5. Must have minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air

Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection
2. Any active, uncontrolled infection.
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
4. Clinically apparent arrhythmia or arrhythmias that are not stable on medical management within two weeks of physician-investigator confirmation of eligibility.
5. Severe, active co-morbidity that, in the opinion of the physician-investigator, would preclude participation in this study.
6. Active acute or chronic GVHD requiring systemic therapy.
7. Dependence on systemic steroids or immunosuppressant medications.
8. Receipt of prior huCART19 or huCART19-IL18 therapy.
9. Active treatment with trimethoprim, methotrexate, or other antifolate chemotherapy, or anticipated use of these drugs during the active treatment phase of the study.
10. Active CNS involvement. Patients with a history of CNS involvement that was successfully treated are eligible. A CNS evaluation is only required for eligibility if a subject is experiencing signs/symptoms of CNS involvement.
11. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
12. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
13. Pregnant or nursing (lactating) patients. Participants of reproductive potential must agree to use acceptable birth control methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2042-09 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor Uptake on [18F]FP-TMP PET/CT | Up to 6 months after huCART19-IL18-eDHFR administration
  In order to evaluate the feasibility of using [18F]FP-TMP PET/CT imaging to detect and measure eDHFR-expressing CAR-T cells, the change in tumor uptake on the post-infusion [18F]FP-TMP PET/CT scans will be compared to baseline.

SECONDARY OUTCOMES:
Evaluate manufacturing feasibility | 3 Months
  The proportion of subjects with huCART19-IL18-eDHFR products that fail to meet the product release criteria, out of the number of eligible subjects in whom manufacturing was attempted,
Incidence of adverse events as assessed by CTCAE v6.0 | up to 15 years after huCART19-IL18-eDHFR administration
  Type, frequency, severity, and attribution of adverse events
Occurrence of Treatment-Limiting Toxicities (TLTs) | 28 days after huCART19-IL18-eDHFR administration
  Unacceptable toxicity as defined by the protocol
Overall Response/Remission Rate (ORR) | Month 3
  Proportion of subjects with CR or PR at Month 3 as compared to baseline
Best Overall Response (BOR) | From Month 3 up to Month 12
  Proportion of subjects with a best overall disease response of CR or PR recorded between the protocol-required Month 3 disease assessment timepoint and the end of primary follow-up (Month 12); or start of new anticancer therapy (including huCART19-IL18-eDHFR retreatment), whichever comes first.
Duration of Response (DOR) | From Month 3 up to 15 years
  Time from the date when the response criteria of CR or PR is first met (at or following Month 3), to the date of confirmed disease progression, death, or other censoring event
Progression-Free Survival (PFS) | Up to 15 years
  Duration of time from huCART19-IL18-eDHFR cell infusion (Day 0) to the date of confirmed disease progression or death.
Overall survival (OS) | Up to 15 years after last huCART-IL18-eDHFR administration
  Duration of time from the first huCART19-IL18-eDHFR infusion (Day 0) to the date of death, for any reason
Retreatment - Overall Response/Remission Rate (ORR) | Up to Month 3-Retreatment
  Proportion of subjects with CR or PR at Month 3-R as compared to retreatment baseline
Retreatment - Best Overall Response (BOR) | From Month 3-Retreatment up to Month 12-Retreatment
  Proportion of subjects with a best overall disease response of CR or PR recorded between the protocol-required Month 3-R disease assessment timepoint and the end of primary retreatment follow-up (Month 12-R); or start of new anticancer therapy, whichever comes first
Retreatment - Duration of Response (DOR) | From Month 3-Retreatment up to 15 years after last huCART-IL18-eDHFR administration
  Time from the date when the response criteria of CR or PR is first met (at or following Month 3-R), to the date of confirmed disease progression, death, or other censoring event
Retreatment - Progression-Free Survival (PFS) | Up to 15 years after last huCART-IL18-eDHFR administration
  Duration of time from huCART19-IL18-eDHFR retreatment infusion (Day 0-R) to the date of confirmed disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schuster, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No